CLINICAL TRIAL: NCT01206985
Title: Pharmacodynamic Study of 125 mg of Paracetamol Permucosal Administered by Sublingual and Buccal Route
Brief Title: Paracétamol PMB by Sublingual et Buccal Routes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Unither SA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CHU-0081; 2010-018746-30 (EudraCT Number)
Record Dates: First submitted 2010-09-06; First posted 2010-09-22 (Estimated); Last update posted 2012-01-30 (Estimated); Status verified 2012-01

CONDITIONS: Healthy Volunteers
Keywords: Paracetamol; per-oral mucosa PMB; No disease, healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider

INTERVENTIONS:
Other: Von Frey electronic — Change in pain threshold testing mechanical stimulation (von Frey electronic)

SUMMARY:
Paracetamol is the analgesic most used, indicated in the symptomatic treatment of fever and pain of mild to moderate. It comes in different dosage forms intended for oral, intravenous and rectal.

The per-oral mucosal route is not used for the administration of paracetamol. It is a very interesting way for the rapid absorption of drugs such as nitrates used in angina pectoris, as it seeks a highly vascular area (the floor of the tongue or gingival groove) and allows very rapid action. In addition, the oral administration-oral mucosa, less restrictive than IV administration and faster than oral administration, seek a single medical procedure unattended after dosing, will entail no pain or risk for infections the patient (in contrast to the IV). The investigators tested a new oral dosage form permucosal (at 250mg/ml) of paracetamol and compared at pharmacological (pharmacokinetic and pharmacodynamic) with the only dosage form of reference used by the IV route in the protocol "Pilot study Pharmacology paracetamol administered oral permucosal PMB. It seems interesting now to reduce the dose by half permucosal to assess how changing the pharmacodynamics of the form permucosal to 125mg/ml. This form will be administered in oral permucosal buccal as well as sublingual (under the pillar of the language) and compared with paracetamol in IV.

DETAILED DESCRIPTION:
Crossover study, double-blind, randomized, controlled versus placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers.
* Aged over 18 years and not more than 50 years.
* Males or female
* Values of vital signs before administration of the test products:
* PAS between 100-140 mm Hg
* PAD between 50-90 mm Hg
* Radial pulse between 45-90 beats per minute
* Free from any treatment in the 7 days preceding inclusion including no use of analgesics or anti-inflammatories

Exclusion Criteria:

* Contraindications to the administration of paracetamol
* Medical history and / or surgical judged by the investigator or his representative as being incompatible with the test, especially subjects with neuropathic pain
* Pathology evolutionary time of the review for inclusion.
* Binge drinking, smoking (more than 10 cigarettes / day), coffee, tea or drinks containing caffeine (equivalent to more than 4 cups per day) or drug abuse.
* Subject does not meet the selection criteria regarding their ability to discriminate the sensations resulting from noxious stimuli during psychometric testing.
* Topic having all breaches of the oral mucosa (aphtes. ..).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Change in pain threshold testing mechanical stimulation (von Frey electronic) | T0-5min, T0+3min, T0+7min, T0+15min, T0+30min, T0+50min, T0+90min

SECONDARY OUTCOMES:
Evaluation of the acceptability of the permucosal product by the subject (evaluation questionnaire). | T0+70min
Analysing a Sample of saliva for enzymatic determination (pharmacogenomics analysis) | T0-10min

CONTACTS AND LOCATIONS:
Overall Officials: Gisèle PICKERING, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France